CLINICAL TRIAL: NCT00204750
Title: A Randomized, Prospective Trial of Electrosurgical Incision Followed by Rabeprazole Versus Bougie Dilation Followed by Rabeprazole of Symptomatic Lower Esophageal (Schatzki's) Rings
Brief Title: Trial of Electrosurgical Incision Versus Bougie Dilation of Symptomatic Lower Esophageal (Schatzki's) Rings
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: University of Utah, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8953
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Lower Esophageal Ring; Dysphagia
Keywords: lower esophageal ring; dysphagia; electrosurgical incision; bougie dilation; GERD
MeSH Terms: conditions — Esophageal Ring, Lower; Deglutition Disorders; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bougie dilation
  Interventions: Procedure: Bougie Dilation
- 2 (Experimental): Needle-knife incision
  Interventions: Procedure: Needle-knife incision

INTERVENTIONS:
Procedure: Bougie Dilation — Bougie dilation will be performed as standard
  Other Names: Maloney dilation
  Arms: 1
Procedure: Needle-knife incision — Needle-knife incision will be performed
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the efficacy of bougie dilation to electrosurgical incision of symptomatic schatzki's rings at one year follow-up in the presence of rabeprazole treatment. All patients will be followed for one year for recurrence and/or severity of dysphagia and will be placed on rabeprazole for that time period.

DETAILED DESCRIPTION:
Fifty consecutive patients referred for endoscopic evaluation at endoscopy labs at the University of Utah Health Sciences Center and the Salt Lake City VA Medical Center for dysphagia will be enrolled in the study prior to endoscopy. If a Schatzki's Ring is found at endoscopy, the patient will be randomized to electrosurgical incision or standard bougie dilation. Patients will be placed on rabeprazole for one year. Follow-up on recurrence and/or severity of dysphagia will be analyzed at interim time periods (1,3,6, 9 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80 with symptomatic Schatzki's ring
* No history of bleeding diathesis or other contraindication to bougie dilation or electrosurgical incision

Exclusion Criteria:

* Contraindication to proton pump inhibitors
* Pregnancy
* Inability to provide informed consent
* History of previous esophagogastric surgery
* Presence of esophageal peptic stricture, esophageal motility disorder or esophageal cancer that could otherwise account for dysphagia
* Nasopharyngeal lesion or nasal intubation intolerance causing inability to undergo esophageal motility testing and ambulatory pH monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Recurrence at one year of Schatzki's ring | One year

SECONDARY OUTCOMES:
GERD score at 1,3,6,9,12 month time intervals | one year
Dysphagia score at 1,3,6,9,12 month time intervals | one year

CONTACTS AND LOCATIONS:
Overall Officials: John Fang, M.D., Study Director — University of Utah HSC; James A DiSario, M.D., Principal Investigator — University of Utah HSC
Locations (1):
- University of Utah HSC, Salt Lake City, Utah, United States